CLINICAL TRIAL: NCT04222660
Title: Diabetic Neuropathy: Function-Structure of Corneal Nerves to Assess Injury-Repair
Brief Title: Corneal Nerves Function and Structure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C0889-R; RX000889-06 (Other Grant/Funding Number: Veterans Adminstration); 5R01DK107399-04 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2020-01-10 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetes; neuropathy; fish oil; cornea; omega 3 polyunsaturated fatty acids
MeSH Terms: conditions — Diabetes Mellitus; Corneal Diseases | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: The study will be done in two phases. In the second phase the investigators will investigate whether increased intake of fish oil improves diabetic peripheral neuropathy including improvement in corneal nerve morphology and sensitivity. Subjects will receive 4g (2g twice a day) of fish oil per day in capsule form. The second phase of the study will be done in 2 of the 3 groups. The two groups for this phase of the study will be the control subjects and the diabetic subjects with neuropathy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Type 2 diabetes without neuropathy (Experimental): Subjects with type 2 diabetes will be enrolled and determination if they have neuropathy will be determined from their clinical record and evaluation.
  Interventions: Dietary Supplement: Blackmores Omega Daily (4 1g capsules per day)
- Type 2 diabetes with neuropathy (Experimental): Subjects with type 2 diabetes will be enrolled and determination if they have neuropathy will be determined from their clinical record and evaluation.
  Interventions: Dietary Supplement: Blackmores Omega Daily (4 1g capsules per day)
- Normal subjects, aged match with no symptoms of diabetes (Experimental): Healthy, aged matched control subjects will be enrolled and determination if they have neuropathy will be determined from their clinical record and evaluation.
  Interventions: Dietary Supplement: Blackmores Omega Daily (4 1g capsules per day)

INTERVENTIONS:
Dietary Supplement: Blackmores Omega Daily (4 1g capsules per day) — Subjects enrolled in phase two of the study will be instructed to take 4 capsules per day (2 in the morning and 2 in the evening). Each capsule contains 1000 mg of triglyceride; 35% eicosapentaenoic acid and 25% docosahexaenoic acid.
  Other Names: fish oil

SUMMARY:
Peripheral neuropathy affects about 50% of the diabetic population and there is no treatment other than good blood glucose control, which is ineffective in subjects with type 2 diabetes. Part of the problem for the lack of an effective treatment is the inability to detect peripheral neuropathy in its early stage. The hypotheses to be addressed in the first phase of this study is that changes in cornea sensitivity (blinking and squinting) following addition of a hyperosmotic solution will provide a novel screening tool for early diagnosis of peripheral neuropathy. For the second phase of the study the investigators will examine the effect of fish oil treatment of diabetic subjects with neuropathy on corneal nerve density and sensitivity. Corneal nerves are the most highly innervated part of the human body with great sensitivity. The first phase will use this property and determine whether sensitivity is lost in diabetic patients with neuropathy. Preclinical studies have supported this hypothesis and now this will be tested in human subjects. Preclinical studies have also shown that treating diabetic rodents with fish oil improves nerve regeneration and outcome measures of peripheral in diabetic rodents. In the second phase the investigators will perform preliminary studies in human subjects with diabetic neuropathy and determine whether treating them with fish oil increases corneal nerve density and sensitivity.

DETAILED DESCRIPTION:
Recruitment has been suspended because of the COVID-19 crisis and the Iowa City VA is just beginning to have face to face appointments.

The hypotheses to be studied in the following specific aims is that changes in cornea sensitivity to a hyperosmotic solution will provide a novel screening tool for early diagnosis of diabetic peripheral neuropathy. The investigators also propose that clinical feasibility studies will demonstrate that treatment with fish oil will improve outcome measures of diabetic peripheral neuropathy.

Specific aims:

1. Determine if the reflex squinting and blinking response to the application of a hyperosmotic solution to the cornea is impaired in patients with type 2 diabetes with or without peripheral neuropathy.

   a. Determine whether changes in corneal sensitivity correlate with loss of cornea nerves in the sub-epithelial layer of the cornea and symptom scores for PN.
2. Determine if treating human subjects with type 2 diabetic peripheral neuropathy with an oral fish oil supplement increases circulating levels of resolvin D1, restores cornea sensitivity to a hyperosmotic eye drop challenge and improves corneal nerve density and symptom scores for peripheral neuropathy.

For this first phase the investigators will enroll 75 subjects to participate (Fifty subjects with type 2 diabetes; 25 with clinically detectable peripheral neuropathy and 25 without neuropathy will be enrolled as well as 25 age-matched control subjects). In the second phase of the study the investigators will investigate whether increased intake of fish oil improves diabetic peripheral neuropathy. Subjects will receive 4g (2g twice a day) of fish oil per day in capsule form.

The investigators first introduced fish oil as a successful treatment of peripheral neuropathy in pre-clinical studies with diabetic rodents and will now expand those studies , culminating in this feasibility study of treatment using human subjects with type 2 diabetes and neuropathy. In this study non diabetic subjects (control) and subjects with type 2 diabetes with mild to moderate peripheral neuropathy will be recruited from phase 1 of this study to participate in the phase 2 treatment phase of the study. A baseline determination of their neuropathy (Subjective Peripheral Neuropathy Screen Questionnaire) including evaluation of corneal nerve structure and sensitivity and blood sample will be performed. Tests besides the questionnaire to be used to screen the subjects for peripheral neuropathy will include 10 g mono filament, vibration threshold, ankle reflex and sensitivity to warm and cold stimulus. Subjects will then be instructed to take 2 fish oil capsules twice a day. Subjects will return at 4, 8 and 12 months for re-evaluation. If successful, the feasibility study will provide a proof of concept to advance fish oils to a larger clinical trial for diabetic peripheral neuropathy.

Visual acuity (subject's vision) will be measured by having the subject read the smallest letters on an eye chart with their glasses or best correction. This takes about 5 minutes or less.

Slit lamp examination: A standard slit lamp examination will be performed to insure that no exclusion criteria are present and no corneal abrasion is present.

The corneal sensitivity procedure will consist of applying a drop of 5% Muro 128 to the eye and recording the blinking and squinting response over the next 5 minutes. Based on preclinical studies it is anticipated that normal subjects will have an increased blinking and squinting response seconds after the addition of the hyperosmotic solution (5% Muro 128), whereas diabetic subjects with neuropathy will have a attenuated response.

Corneal sensation threshold: Corneal sensation will also be measured in each eye using a handheld Luneau Cochet -Bonnet aesthesiometer. This device contains a thin, retractable, nylon monofilament in which the length (stiffness) is varied between 6.0 mm and 1.0 mm until the subject can detect the touch on their central cornea, resulting in a blink reflex. In each eye, testing will begin with the 6.0 mm filament, after which the length will be progressively shortened by 0.5 mm until the patient reports sensing the corneal contact. Each eye will be tested three times and the best performance (in terms of longest filament that is perceived to touch the cornea) will be recorded as the corneal sensation threshold.

Ocular Coherence Tomography (OCT):

The thickness of the optic nerve and macula will also be measured inside of the eye using a special camera that forms an image of the layers of the retina. The imaging is harmless and measures the thickness or structural health of retinal layers and optic nerve. A new feature of OCT is eye-tracking. Eye tracking does not take any longer since it is done simultaneously with the imaging. Eye tracking during OCT may give us new insight into some eye disorders. This test takes approximately 10 minutes.

A hand-held pupillometer/electroretinogram device (RETeval, LKC) will be held in front of the subject s eye, but will not touch the eye. The device will provide a brief, a series of brief light stimuli and then record the pupil response and the elicited electrical response from the retina from a surface skin patch (electrode) placed below each eye, from the light as a measure of whether the inherent sensitivity of the eye in the retina is normal. The investigators will repeat this in the left eye. The visible light stimulus is safe and is given at an intensity experienced in normal daily light exposures. The test takes about 2 minutes per eye.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients diagnosed based on the opinion of an Endocrinologist (Dr. Correia), the absence of a history of ketoacidosis, and a C-peptide > 0.8 ng/ml
* At least 5 year known duration of diabetes.
* HbA1c < 9.0%
* None or mild to moderate peripheral neuropathy based on medical record, Michigan Neuropathy Screening Instrument including response to monofilament test, ankle reflex test, vibration perception threshold examination using a 128 Hz tuning fork as well as hot and cold sensation evaluation

Exclusion Criteria:

* Any neurologic, muscular, genetic, or other condition known to affect nerve or muscle function
* Electrolyte abnormalities, untreated hypothyroidism, abnormalities in calcium, phosphate, or magnesium concentrations, or any other metabolic disturbance affecting neural function
* Cigarette smoking in the past year
* Peripheral vascular, cardiac, pulmonary, or any other disorder affecting blood or tissue oxygenation
* Risk of bleeding disorder or on medication known to increase risk of bleeding
* History for use of aspirin
* Any other medical or psychological condition judged to limit compliance with the protocol or interpretation of results
* History of diabetic foot ulcer
* LDL > 100 mg/100ml, HDL < 30 mg/100ml, Triglyceride > 400 mg/100ml.* 10) BP < 140 systolic and 80 diastolic
* BMI 45
* Insulin use to manage diabetes 200 units
* History of taking fish oil supplements
* The investigators are limiting subject population to those over 50 thus pregnancy should not be an issue nonetheless females who are pregnant, looking to become pregnant or are breast feeding will be excluded (* After overnight fast of 8-12 h; Average of three determinations in the sitting position after at least 5 minutes rest.)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2025-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Yorek, PhD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reviewer is correct. Due to the pandemic the course of this study was dramatically changed. Initially there was going to be 2 separate protocols the first to measure cornea sensitivity using a hyperosmotic solution in 3 groups control, and diabetes with or without neuropathy. The second protocol was to be treatment with fish oil to determine whether improvement occurs. Because of COVID we were able to complete only protocol 1 and it was done in only control and diabetes neuropathy subjects.
Period: Overall Study
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Started | 28 | 16
Completed | 28 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes | Total
Number analyzed (Participants) | 28 | 16 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 15 | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (1.9) | 49.8 (5.0) | 56.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 24 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 26 | 15 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 24 | 15 | 39
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 16 | 44
cornea sensitivity using isotonic solution [Mean (Standard Deviation); unit: time ratio eyelids closed vs. open] | 0.089 (0.012) | 0.085 (0.027) | 0.088 (0.010)
cornea sensitivity using Cochet-Bonnet [Mean (Standard Deviation); unit: cm] | 5.68 (0.47) | 5.95 (0.14) | 5.78 (0.41)
nerve conduction [Mean (Standard Deviation); unit: m/s] | 35.6 (13.2) | 50.5 (10.4) | 41.0 (13.4)
nerve amplitude [Mean (Standard Deviation); unit: uV] | 3.80 (1.39) | 14.63 (6.86) | 7.74 (6.98)
Dry eye (DEQ 5) questionnaire [Mean (Standard Deviation); unit: units on a scale] — The minimum is 0 (healthy) to 22 (extremely poor)
  units on a scale | 7.12 (5.30) | 2.00 (3.31) | 5.26 (5.31)
Ocular Surface Disease Index (OSDI) questionnaire [Mean (Standard Deviation); unit: units on a scale] — Based on their OSDI scores, patients can be categorized as having a normal ocular surface (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) ocular surface disease. Full scale is 0 - 100.
  units on a scale | 11.36 (9.80) | 1.09 (2.59) | 7.63 (9.20)
Michigan neuropathy screening instrument [Mean (Standard Deviation); unit: units on a scale] — The scale for this test ranges from 0 (healthy) to 13 (poor). A value above 4 indicates presence of peripheral neuropathy.
  units on a scale | 5.72 (2.52) | 0.54 (1.03) | 3.84 (3.68)

OUTCOME MEASURES:

1. Primary Outcome: Cornea Sensitivity
Description: Cornea sensitivity to a isotonic and hyperosmotic solution is evaluated as the amount of time the eyelid is closed over a period of 150 seconds following application of first isotonic saline (0.9% NaCl) followed by Muro 128 (5% NaCl solution) after a 5 minute recovery/washout period. The evaluation is done from analyzing the recordings of each event using a multi-camera video platform. The results are reported for response to saline (baseline) and Muro (stimulant) solutions as a ratio of the time the eyelids are closed vs. open over the 150 second period of the recording.
Time Frame: Examination of the response to saline and Muro 128 is preformed once in each patient immediately following their consent or if they request at a later more convenient time.
Population: primary outcome
Measure: Mean (Standard Deviation); unit: time ratio of eyelids closed vs. open
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
time ratio of eyelids closed vs. open | 0.177 (0.073) | 0.293 (0.036)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.001, ANOVA

2. Secondary Outcome: Change in Corneal Sensation Threshold Using Cochet Bonnet Filament
Description: This test records the mechanical sensitivity of the cornea to a filament that is touched to the cornea. The rigidity of the filament can be adjusted and the outcome is the length of the filament (6 to 1 cm) when the subjects blinks. The data will be recorded as cm.
Time Frame: Done once to determine whether there is a difference between control and diabetes subjects with peripheral neuropathy
Measure: Mean (Standard Error); unit: cm
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
cm | 5.683 (0.066) | 5.953 (0.026)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0025, t-test, 2 sided

3. Secondary Outcome: Michigan Neuropathy Screening Instrument
Description: All subjects will answer a 15 question survey that relates to symptoms of peripheral neuropathy. The score range is 0-13 with the higher score indicating poorer outcome or increased peripheral neuropathy.
Time Frame: Done once as part of the determination to the subjects peripheral neuropathy.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
units on a scale | 5.720 (0.0505) | 0.5455 (0.3123)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Sensitivity to 10 g Monofilament Test
Description: The 10 g monofilament test is a routine evaluation used to screen the diabetic foot for loss of sensory sensation and part of the standard of care for any diabetic patient. The subject will remove their footwear and lie down on a table. The filament will be applied perpendicular to the skin surface on the bottom of the feet will sufficient force to allow the filament to bend. This is repeated 5 times. Each subject will be asked to tell the examiner if they feel it. The scale is 0 to 1. If the subject feels the monofilament the value each time the score given is 0. If there is no feeling the value is 1. For reduced sensitivity, for example feels the monofilament 2 or 3 times during the test the score is 0.5. A higher score is evidence of peripheral neuropathy.
Time Frame: Done once as a determination of the presence of peripheral neuropathy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
units on a scale | 0.5577 (0.07507) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Presence of Vibratory Sensation of the Great Toe
Description: Vibratory sensation is a standard of care test used with patients with diabetes to test sensory nerve sensation. A 128 Hz tuning fork is used and placed over the dorsum of the great toe on the boney prominence of the distal interphalangeal joint. The subject is asked to tell the examiner if they feel the object touching their toe. This is repeated 3 times. The scale is 0 to 1. If the subject feels the object the score given is 0. If the subject fails to feel the object all 3 times the score is 1. If they feel it once or twice during the examination the score given is 0.5. A higher score is evidence of peripheral neuropathy.
Time Frame: Done once as a determination of the presence of peripheral neuropathy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
units on a scale | 0.6731 (0.0551) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Presence of Reflex
Description: Reflex testing is commonly used to detect sensory neuropathy in diabetic patients. The ankle reflex is examined by aligning the subjects ankle into a neutral position and the examiner strikes the Achilles tendon with a neurological hammer. An abnormal result is recorded if the subject does not display any ankle plantarflexion. The scale is 0 to 1. If the reflex is present the score given is 0. If no reflex is present the score given is 1. If the response is reduced the score given is 0.5. A higher score is evidence of peripheral neuropathy.
Time Frame: Done once as a determination of the presence of peripheral neuropathy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
units on a scale | 0.8125 (0.07855) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0001, t-test, 2 sided

7. Secondary Outcome: Visual Acuity
Description: A routine visual acuity eye examination will be performed. Subjects vision will be measured by having the subject read the smallest letters on an eye chart with their glasses or best correction.
  Visual acuity (VA) is a measure of the ability of the eye to distinguish shapes and the details of objects at a given distance (20 feet). A person with "normal vision" scores 20/20 as did all our controls. A person with 20/40 vision sees things at 20 feet that most people who don't need vision correction can see at 40 feet. Our subjects with diabetic neuropathy mean score was 20/25. The first number in the score is the number of feet for the test and this is commonly 20 feet. The second number is their visualization of the letters on the eye chart. The investigators used the mean of the second number for analysis. This takes about 5 minutes or less.
Time Frame: Done once to determine the subjects visual ability
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
units on a scale | 25 (0.001) | 20 (0.000)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.01, t-test, 2 sided

8. Secondary Outcome: Questionnaires for Corneal Sensitivity
Description: Ocular Surface Disease Index (OSDI contains 12 questions relating to eye sensitivity to light, vision acuity, dryness, sensitivity when reading, using the computer, and watching TV). The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability.
Time Frame: Done once to determine extent of common eye disease such as dry eye
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
units on a scale | 11.36 (1.96) | 1.09 (0.78)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0017, t-test, 2 sided

9. Secondary Outcome: Determination of Tibial Nerve Conduction Velocity
Description: This is a non-invasive method of determining conduction velocity of the tibial nerve. the scale is meters per second or m/s. The subject will be instructed to lie down on a examination table with shoes and socks removed. Afterwards, the lower ankle will be swabbed with an alcohol patch and allowed to air dry. A device containing 2 posts (about 3 inches apart) will be placed on the lower ankle in the region of the Achilles and activated. For a period of 5-10 sec the device sends a pulse stimulating the nerve distally (post located at the lower part of the ankle) and the response recorded by the post located distally on the skin of the upper part of the ankle. The nerve conduction is recorded electronically by the device and data down loaded to a secured computer. During the time of the analyses the subject will feel dual pulsating sensation that will last up to 10 sec.
Time Frame: Done once as a determination of the presence of peripheral neuropathy
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
Number analyzed (Participants) | 28 | 16
m/s | 35.60 (4.19) | 50.50 (3.68)
Statistical Analysis 1: Comparison: Type 2 Diabetes With Neuropathy vs Normal Subjects, Aged Match With no Symptoms of Diabetes; Test type: Other; p < 0.0195, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The procedure for each subject lasted a total of no more than 2 hours. None of the procedures were invasive and had very low risks. The subject was monitored during the procedures.
Description: The only possible adverse event would have been eye discomfort due to the Muro 128 solution. However, after this procedure the subjects eyes were flushed with warm saline. The total time each participant took to complete the study was 2 hours. For this reason all-cause mortality was not monitored.
Arm/Group | Type 2 Diabetes With Neuropathy | Normal Subjects, Aged Match With no Symptoms of Diabetes
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/16
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

LIMITATIONS AND CAVEATS:
Study weaknesses include the number of subjects enrolled being primarily male. The control group was not well age matched. Recruitment of diabetes subjects was restricted to those with known peripheral neuropathy. Additional studies are needed that include diabetes subjects without peripheral neuropathy and those with mild peripheral neuropathy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT04222660/Prot_SAP_000.pdf